CLINICAL TRIAL: NCT01813474
Title: A Phase I, Open-label Study to Assess the Safety and Tolerability of Doses of Olaparib Tablet in Japanese Patients With Advanced Solid Malignancies
Brief Title: Investigate the Safety and Tolerability of Olaparib Tablet in Japanese Patients With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D081BC00001
Record Dates: First submitted 2013-03-15; First posted 2013-03-19 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-01-16 (Actual); Status verified 2017-12

CONDITIONS: Cancer; Advanced Solid Malignancies
Keywords: Cancer; Tumour; Solid Malignancies
MeSH Terms: conditions — Neoplasms | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- olaparib tablet monotherapy (Experimental): olaparib tablet
  Interventions: Drug: olaparib

INTERVENTIONS:
Drug: olaparib — tablet oral

SUMMARY:
The objective of this study will be to investigate the safety and tolerability of olaparib tablet when given orally to Japanese patients with advanced solid malignancies. In addition, the pharmacokinetic profile, MTD (if possible) and efficacy of olaparib will be investigated.

DETAILED DESCRIPTION:
MTD - maximum tolerated dose

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with advanced solid malignancies who are refractory to standard therapies or for which no standard therapy exists.
* Subjects who have overall good overall general condition.
* Subjects who agree to hospitalisation from starting olaparib to multiple dose period at day 15.
* Evidence of non-childbearing status for women of childbearing potential, or postmenopausal status.
* Subjects who have at least one lesion (measurable and/or non-measurable) that can be accurately assessed by CT/MRI at baseline and follow up visits

Exclusion Criteria:

* Subjects who received any previous treatment with a PARP (poly adenosine diphosphate-ribose polymerase) inhibitor, including olaparib.
* Subjects receiving inhibitors of CYP3A4 (cytochrome P450 3A4).
* Subjects with symptomatic uncontrolled brain metastases.
* Subjects with myelodysplastic syndrome/acute myeloid leukaemia.
* Subjects with a known hypersensitivity to olaparib or any of the excipients of the product.

Ages: 20 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-03-25 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Morris, M.D., Study Director — Global Medicines Development
Locations (3):
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Sapporo

REFERENCES:
- See also: D081BC00001_Study_Report_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1680&filename=D081BC00001_Synopsis.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 25 March 2013. Last patient enrolled on 31 October 2013. Data cut off on 31 July 2014.
Pre-assignment Details: A total of 28 participants gave informed consent to join this study. Five participants were screen failures so that 23 participants were assigned and received study treatment
Groups:
- 200 mg Bid, Dose Escalation Part: Olaparib tablet 200 mg bid, 400 mg/day, dose escalation part
- 300 mg Bid, Dose Escalation Part: Olaparib table 300 mg bid, 600 mg/day, dose escalation part
- 300 mg Bid, Expansion Part: Olaparib tablet 300 mg bid, 600 mg/day, expansion part
Period: Overall Study
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part | 300 mg Bid, Expansion Part
Started | 4 | 7 | 12
Completed | 1 (ongoing study at final data cut off) | 0 | 1 (ongoing study at final data cut off)
Not Completed | 3 | 7 | 11
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lack of Efficacy | 2 | 6 | 9
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part | 300 mg Bid, Expansion Part | Total
Number analyzed (Participants) | 4 | 7 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.0 (8.68) | 55.4 (8.98) | 57.3 (12.43) | 54.1 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 4 | 4 | 7 | 15
  Sex: Male | 0 | 3 | 5 | 8
Primary tumour location [Count of Participants; unit: Participants]
  Breast | 1 | 1 | 3 | 5
  Colorectal | 0 | 0 | 1 | 1
  Lung | 0 | 1 | 2 | 3
  Peritoneum | 0 | 0 | 1 | 1
  Pancreas | 0 | 1 | 0 | 1
  Ovary | 0 | 2 | 2 | 4
  Uterus | 1 | 1 | 0 | 2
  Cervix | 2 | 0 | 0 | 2
  Colon | 0 | 0 | 1 | 1
  Gastric Antrum | 0 | 0 | 1 | 1
  Other | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. This was recorded if it happend from the start dose to 30 days after the last of study drug.
Time Frame: From the start dose to 30 days after the last dose of study drug
Measure: Number; unit: Participants
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part | 300 mg Bid, Expansion Part
Number analyzed (Participants) | 4 | 7 | 12
Participants
  At least 1 Adverse Events (AE) | 4 | 7 | 10
  At least 1 AE of CTCAE Grade 3 or higher | 1 | 3 | 1
  At least 1 Serious Adverse Events (SAE) | 1 | 0 | 0

2. Secondary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Dose Limiting Toxicities were defined as study specific events that is determined to be possibly or probably related to olaparib (as determined by the investigator) and occurring during the first cycle of treatment (28 days after the first dose), irrespective of whether the toxicity resolved.
Time Frame: From the start dose to 28 days after the first dose of study drug
Population: All patients in only the dose escalation part who received olaparib and completed the safety follow-up through the dose-limiting toxicity (DLT) evaluation period (28 days), or who experienced a DLT.
Measure: Number; unit: Participants
Groups:
- 300 mg Bid, Dose Escalation Part: Olaparib tablet 300 mg bid, 600 mg/day, dose escalation part
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

3. Secondary Outcome: Cmax Following Single Dosing
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours at post-dose
Population: Dose escalation part only
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part
Number analyzed (Participants) | 4 | 7
μg/mL | 6.697 (95.69) | 7.743 (34.76)

4. Secondary Outcome: Cmax Following Multiple Dosing
Time Frame: Day 15: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours at post-dose
Population: Dose escalation part only. Two participants (1 in 200 mg bid and 1 in 300 mg bid) had no PK data due to early discontinuation prior to Day 15.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part
Number analyzed (Participants) | 3 | 6
μg/mL | 7.668 (46.93) | 8.434 (35.05)

5. Secondary Outcome: Tmax Following Single Dosing
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours at post-dose
Population: Dose escalation part only
Measure: Median (Full Range); unit: hour
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part
Number analyzed (Participants) | 4 | 7
hour | 2.00 (95.69) [1.00 to 3.00] | 1.98 (34.76) [1.00 to 3.00]

6. Secondary Outcome: Tmax Following Multiple Dosing
Time Frame: Day 15: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours at post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part
Number analyzed (Participants) | 3 | 6
hour | 1.50 (46.93) [1.00 to 3.00] | 3.00 (35.05) [1.50 to 3.93]

7. Secondary Outcome: AUC Following Single Dosing
Time Frame: Day 1: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48 hours at post-dose
Population: Dose escalation part only. One participant in 200 mg bid had no AUC data because AUC was not calculable for this participant.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part
Number analyzed (Participants) | 3 | 7
μg*h/mL | 61.97 (473.4) | 46.21 (64.64)

8. Secondary Outcome: AUC at Steady State Following Multiple Dosing
Time Frame: Day 15: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hours at post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part
Number analyzed (Participants) | 3 | 6
μg*h/mL | 36.50 (71.94) | 52.34 (68.17)

ADVERSE EVENTS:
Time Frame: Through treatment and 30-day follow-up period, an average of about 4 months.
Arm/Group | 200 mg Bid, Dose Escalation Part | 300 mg Bid, Dose Escalation Part | 300 mg Bid, Expansion Part
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/7 | 0/12
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 10/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg Bid, Dose Escalation Part (N=4) | 300 mg Bid, Dose Escalation Part (N=7) | 300 mg Bid, Expansion Part (N=12)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 200 mg Bid, Dose Escalation Part (N=4) | 300 mg Bid, Dose Escalation Part (N=7) | 300 mg Bid, Expansion Part (N=12)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dysaesthesia pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 6 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 2
Malaise (General disorders) | 0 | 2 | 2
Oedema (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 1
Grip strength decreased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 2 | 2
Platelet count decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No